CLINICAL TRIAL: NCT01185028
Title: An Open-Label Safety and Tolerability Study of Nitazoxanide, Pegylated-Interferon Alfa 2a and Ribavirin in HIV/HCV Co-Infected Genotype 1 Prior Treatment Relapsers and Non-Responders
Brief Title: A Safety and Tolerability Study of Nitazoxanide in HIV-HCV Treatment Failures
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100183; 10-CC-0183
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Results first posted 2013-05-15 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2013-05

CONDITIONS: Hepatitis C Infection; HIV Infection
Keywords: Chronic HCV; HCV Treatment Nonresponders; HCV Treatment Relapsers; HIV-HCV Co-Infection; Nitazoxanide; Hepatitis C
MeSH Terms: conditions — Hepatitis C; HIV Infections | interventions — nitazoxanide; Ribavirin

ARMS (1):
- Nitazoxanide With Pegylated Interferon And Ribavirin (Experimental): Nitazoxanide 500mg po bid for 4 wks followed by peg-IFN/Ribavirin/nitazoxanide for 48 weeks
  Interventions: Drug: Nitazoxanide With Pegylated Interferon And Ribavirin

INTERVENTIONS:
Drug: Nitazoxanide With Pegylated Interferon And Ribavirin — Nitazoxanide 500mg po bid for 4 wks followed by peg-IFN/Ribavirin/nitazoxanide for 48 weeks

SUMMARY:
Background:

* Chronic hepatitis C (CHC) is a major health problem that particularly affects individuals with human immunodeficiency virus (HIV) infection, and can lead to cirrhosis and liver failure. Standard treatment for people with HIV and CHC is a 48-week course of pegylated-interferon alfa 2a (peg-IFN) and ribavirin (RBV), but better treatments are needed for those who either do not respond to the drugs or who relapse after treatment.
* Nitazoxanide has been approved by the Food and Drug Administration primarily to treat diarrhea caused by parasites, and it has been studied in the treatment of CHC infection. However, it has not been tested in persons infected with HIV and CHC co-infection. Researchers are interested in determining whether nitazoxanide is a safe and tolerable treatment for CHC in individuals with HIV.

Objectives:

- To assess the safety and tolerability of using nitazoxanide to treat chronic hepatitis C infection in individuals with HIV who have not responded to standard treatment for hepatitis C.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with both HIV and chronic hepatitis C, and who have either not responded to or relapsed after previous hepatitis C treatment.

Design:

* Participants will be screened with a physical examination and medical history; blood and urine tests; imaging studies; possible heart, lung, and psychological tests; and a liver biopsy if one has not been done in the past 3 years.
* Participants will receive nitazoxanide, the medication being studied, to take by mouth for 4 weeks, and will provide blood samples during this time.
* After 4 weeks, participants will receive the first dose of peg-IFN and RBV. Participants will have weekly injections of peg-IFN and continue to take nitazoxanide and RBV by mouth for 48 weeks. Individuals who are slow to respond to this combined CHC treatment (nitazoxanide, peg-IFN, and RBV) by week 12 will continue to have the combined treatment for an extended period, a total of 72 weeks.
* Participants will have study visits to provide blood samples and have other tests two times in the first month of combined treatment, and then at months 2, 3, 4, 7, 10, 13, 19; and month 25 only in participants slow to respond to combined treatment.
* Some participants who are on specific HIV treatment regimens may enroll in a substudy that will require three separate 12-hour visits for repeated blood samples and other tests during the initial 4-week nitazoxanide treatment.

DETAILED DESCRIPTION:
Chronic hepatitis C (CHC) viral infection is a major health problem affecting 130-170 million worldwide, and 2.7-3.9 million in the US, more than 3 times those with HIV infection. One-third of persons with HIV have CHC, a more rapid progression to cirrhosis and liver failure, with liver disease as one of the leading causes of mortality.

Standard treatment, pegylated-interferon (IFN) alfa and ribavirin (RBV), has an efficacy, sustained virologic response (SVR), of less than 50% in those with HCV genotype 1 (GT 1); and only about 25% of those with HIV-HCV GT1 co-infection. SVR is even lower in those retreated, who were prior treatment relapsers or non-responders; few published studies exist, especially in those with HIV. Improved therapy is imperative given increasing morbidity and mortality and the proportion of persons who are relapsers or non-responders. Newer and promising anti-HCV therapies, directly acting antivirals (DAA), are in development. However, only 2 are in Phase 3 clinical trials and most remain far from FDA approval.

An oral agent, nitazoxanide (NTZ), with broad in vitro anti-microbial activity and a good safety profile, has higher efficacy rates in treatment na ve participants mono-infected with HCV GT 1 or 4. There have not been studies in HIV co-infected persons, nor pharmacokinetic (PK) studies in liver or renal disease. In vitro studies suggest that NTZ has both a direct suppressive effect on HCV replication, as well as a sensitizing effect on IFN-mediated suppression of HCV replication, yet the exact mechanism of action giving rise to higher SVR rates is not well understood.

This is an open-label study in 35 HIV-HCV GT 1 co infected persons, prior relapsers (n=25) or non-responders (n=10) after a full course of IFN and RBV therapy. Participants will receive 4 weeks of NTZ lead-in therapy, followed by NTZ/peg-IFN/RBV triple combination therapy for an additional 48 weeks. Slow responders will receive 72 weeks of triple therapy after the 4-week NTZ lead-in.

The primary endpoint is safety and tolerability of NTZ. Secondary endpoints are exploratory: (1) efficacy rate estimation, (2) viral dynamics assessment, and determination of predictive response, (3) pharmacologic level assessment, (4) indirect mechanistic action evaluation of NTZ through virologic response, and, (5) IFN-stimulated genetic expression evaluation and determination of predictive response. There will be a sub-study evaluating the PK of NTZ in a group of 10 participants who are on a ritonavir-based HIV antiretroviral regimen.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

To be eligible for participation on this protocol, a participant must satisfy all of the following conditions:

Be greater than or equal to 18 years old and have an identifiable Primary Care Provider.

Have either documentation of HIV-1 infection by licensed enzyme-linked immunosorbent assay (ELISA) and confirmed by a Western Blot or HIV RNA of 1,000 copies/mLor greater.

Have documentation of chronic HCV (CHC) infection by demonstration of a positive test for hepatitis C antibocy and HCV RNA of 2,000 IU/mL or greater

Have histopathologic features consisten with CHC at the time of enrollment. A liver biopsy done for a participant with 36 months prior to his or her participant may be used as the baseline biopsy. Participants can opt out of a biopsy if they had one or more than 36 months prior and have a contraindication, sucha as receiving chronic anticoagulation therapy. Participants with decompensated liver disease are excluded from study.

Are co-infected infected with HCV genotype 1 and HIV viruses.

1. Relapsers: Participants who had an undetectable HCV RNA (< 10 IU/mL) at the end of prior treatment (ETR) but have detectable HCV RNA by Week 72 or thereafter.
2. Non-responders: Participants who have received at least 12 weeks of treatment with any IFN alfa 2a or 2b with ribavirin and have not achieved either a 2 log (10) drop in HCV viral levels at week 12 (null responder) nor has not achieved a HCV RNA below the level of detection by Week 24 (< 10 IU/mL).
3. Washout period from prior treatment of at least 3 months.

   Participants with CD(4) cell counts greater than or equal to 100 cells/mm(3)

   Capacity to understand and sign or thumbprint the Informed Consent document, as well as willingness to comply with the study requirements and clinic policies.

   Absolute neutrophil count > 1,000 cells/mm3.

   Platelets > 50,000/mm3.

   Hemoglobin > 10.5 mg/dL.

   Not pregnant or breast-feeding. Serum pregnancy test must be negative 2 weeks prior to Day -28 and to Day 0 prior to dosing with study medications for female participants.

   If the participant is able to become pregnant, then she must use 2 effective methods of contraception during the study. Effective contraceptive methods include abstinence, surgical sterilization of either partner, barrier methods such as diaphragm, condom, cap, or sponge, or use of hormonal contraception with an anti-HIV regimen that will not alter metabolism of hormonal contraception. This is advised on the basis of using ribavirin, which may have a potential teratogenic effect on the fetus in pregnant women. NTZ had not been studied during lactation.

   Be willing to not become pregnant until 6 months after completion of ribavirin therapy.

   Male participants who are not documented to be sterile agree to either abstain from intercourse or consistently and correctly use a condom while their female partner (if applicable) agrees to use one of the appropriate medically accepted methods of birth control listed above from the date of screening until 6 months after their last dose of ribavirin.

   Participants with documented illicit drug use must demonstrate ability to adhere to HIV medication (with an undetectable or stable HIV viral load) and their prior primary care provider appointments (more than 80% as scheduled).

   Be willing to abstain from alcohol use during the trial and enter treatment program if necessary.

   Be able to learn to safely inject medication, be able to find another person or a clinic to inject the medication for him/her, or is willing to come to the clinic for weekly injections.

   Be willing to allow stored blood or tissue samples to be used in the future.

   EXCLUSION CRITERIA

   A participant will be ineligible to participate on this study if any of the following criteria are met:

   A participant cannot be on other experimental therapies (including expanded access/compassionate use of antiretrovirals) for 28 days prior to Day -28 and during his/her participation in this protocol.

   Mixed genotypes (e.g., 1 & 2, 1 & 3,1 & 4). Mixed genotype 1a/1b will be enrolled.

   Has any other known, or clinically suspected, cause of liver disease, including active hepatitis B.

   For participants with cirrhosis, a Child Turcotte Pugh score > 7, or Child's B or C cirrhosis.

   Has a prothrombin time International Normalized Ratio (PT-INR) > 2 and is not on chronic anti-coagulation medications, or has a history of hemophilia.

   Has had an organ transplantation other than cornea or hair.

   Has an estimated creatinine clearance (estimated glomerular flow rate) < 50 mL/min.

   For a participant with higher than 20 ng/mL of alpha-fetoprotein, a negative ultrasound or computerized tomography scan to rule out hepatoma is required for enrollment.

   Has any neoplastic disease EXCEPT for (1) Kaposi's sarcoma not requiring systemic chemotherapy, (2) any non-metastatic skin cancer that has been resected or (3) non-metastatic cervical or anal cancer that has been resected.

   Has evidence of severe cardiac disease (greater than or equal to Grade 3 congestive cardiac failure, symptomatic coronary artery disease, significant arrhythmias, or uncontrolled hypertension) despite intervention or medical therapy.

   Has evidence of severe chronic pulmonary disease with functional impairment or a DLCO (diffusing capacity of the lung for carbon monoxide) less than or equal to 70% at baseline.

   Has a severe psychiatric disorder that would interfere with the adherence to protocol requirements, and that is not stably treated with risk of decompensation.

   Has evidence of autoimmune disorders including inflammatory bowel diseases, psoriasis, and optic neuritis.

   Has evidence of an uncontrolled seizure disorder defined as more than 1 episode of generalized seizure within the past year.

   Has chronic pancreatitis.

   Has severe retinopathy, as determined by the ophthalmologist.

   Has any hemoglobinopathy (e.g., Thalassemia, sickle cell disease).

   Is currently taking didanosine or d4T as part of antiretroviral regimen.

   If total bilirubin is greater than 1.5 mg/dL then direct bilirubin can be no more than 70% of the total, up to a direct bilirubin of 2.0 mg/dL.

   Concurrent use of any immunosuppressive therapy, including systemic steroids (prednisone equivalent of > 10 mg/day) for a duration of 6 weeks or more within 6 months prior to enrollment. Inhaled steroids will be allowed, even with ritonavir.

   Has active systemic infections other than HCV and HIV.

   Has a hepatic mass suggestive of hepatocellular carcinoma as detected by ultrasound scan, dual-phase computerized tomography, or magnetic resonance imaging.

   Has evidence of moderate or heavy alcohol use (> 50 grams/day), or substance abuse, within the past 6 months that potentially could interfere with participant compliance. (Urine toxicology will be completed at screening.)

   Currently uses warfarin, ganciclovir, isoniazid, pyrazinamide, rifabutin, rifampin/rifampicin, thalidomide, or theophylline.

   Has a history of esophageal or gastric varices.

   Has any systemic illness that will make it unlikely that the participant will be able to return for the required study visits.

   Has evidence of gastrointestinal malabsorption, chronic nausea, or vomiting.

   The participant is the male partner of a pregnant woman and does not always use a condom during intercourse.

   Women who are pregnant.

   Women who are breast-feeding.

   Has a hypersensitivity to NTZ, interferon products, or ribavirin.

   Has ingested silymarin (milk thistle), s-adenosylmethionine (SAM-e), glycyrrhizin, Sho-saiko-to (SST), or other herbal supplements that may be either liver beneficial or toxic, within 28 days prior to Day -28.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shyamasundaran Kotilil, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (4):
- United States (4):
  - Family Medical and Counseling Services, SE, Washington D.C., District of Columbia
  - Unity Health Care/Walker Jones, NE, Washington D.C., District of Columbia
  - Whitman Walker Clinic, NW, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Seeff LB, Buskell-Bales Z, Wright EC, Durako SJ, Alter HJ, Iber FL, Hollinger FB, Gitnick G, Knodell RG, Perrillo RP, et al. Long-term mortality after transfusion-associated non-A, non-B hepatitis. The National Heart, Lung, and Blood Institute Study Group. N Engl J Med. 1992 Dec 31;327(27):1906-11. doi: 10.1056/NEJM199212313272703. PMID 1454085
- [Background] Seeff LB. Natural history of chronic hepatitis C. Hepatology. 2002 Nov;36(5 Suppl 1):S35-46. doi: 10.1053/jhep.2002.36806. PMID 12407575
- [Background] Staples CT Jr, Rimland D, Dudas D. Hepatitis C in the HIV (human immunodeficiency virus) Atlanta V.A. (Veterans Affairs Medical Center) Cohort Study (HAVACS): the effect of coinfection on survival. Clin Infect Dis. 1999 Jul;29(1):150-4. doi: 10.1086/520144. PMID 10433578

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitazoxanide With Pegylated Interferon And Ribavirin
Started | 8
Completed | 4
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Nitazoxanide With Pegylated Interferon And Ribavirin
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean has been calculated to the third decimal place. Standard Deviation value has been calculated to the thirteenth decimal place
  years | 56.375 (7.4487834577198)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events determined and evaluated by patient reporting and the DAIDS toxicity table.
Time Frame: 1 year and 2 months
Measure: Number; unit: participants
Arm/Group | Nitazoxanide With Pegylated Interferon And Ribavirin
Number analyzed (Participants) | 8
participants | 8

2. Secondary Outcome: Sustained Viral Response Rate
Description: Proportion of participants that are HCV negative 6 months after treatment completion
Time Frame: 1 year and 2 mos
Measure: Number; unit: participants
Arm/Group | Nitazoxanide With Pegylated Interferon And Ribavirin
Number analyzed (Participants) | 8
participants | 8

3. Secondary Outcome: Tolerability of Study Drug Measured as Discontinuation.
Description: Proportion of individuals that discontinued study drug due to intolerability.
Time Frame: 1 year and 2 mos
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide With Pegylated Interferon And Ribavirin
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Arm/Group | Nitazoxanide With Pegylated Interferon And Ribavirin
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide With Pegylated Interferon And Ribavirin (N=8)
Alanine aminotransferase increased (Investigations) | 1 (9)
Aspartate aminotransferase increased (Investigations) | 1 (14)
Blood glucose increased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (9)
Fatigue (General disorders) | 1 (3)
Blood creatinine increased (Investigations) | 1 (1)
Blood albumin decreased (Investigations) | 1 (8)
Chromaturia (Renal and urinary disorders) | 1 (2)
Blood potassium increased (Investigations) | 1 (1)
Chills (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (3)
Abscess oral (Infections and infestations) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood calcium decreased (Investigations) | 1 (2)
Blood potassium decreased (Investigations) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (10)
Platelet count decreased (Investigations) | 1 (7)
Serum albumin decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes